CLINICAL TRIAL: NCT05345769
Title: A Prospective, Multi-Center, Open-label, Sequential, Multiple Ascending-Dose and High Concentration Cohorts Phase 1 Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Efficacy of AM712 Following Intravitreal Administration in Patients with Neovascular Age-related Macular Degeneration.
Brief Title: Safety and Efficacy of AM712 in Patients with NAMD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AffaMed Therapeutics Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AM712E1001
Record Dates: First submitted 2022-04-12; First posted 2022-04-26 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-11

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: nAMD

STUDY DESIGN:
Masking Description: The Phase 1 study is comprised of open-label multiple ascending-dose component (Part 1) and high concentration component (Part 2) to evaluate the safety, tolerability, pharmacokinetics, and efficacy of AM712 in patients with neovascular age- related macular degeneration (nAMD).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Phase I- All (Experimental): Subjects with neovascular AMD
  Interventions: Biological: AM712(ASKG712)

INTERVENTIONS:
Biological: AM712(ASKG712) — AM712 is a recombinant anti-VEGF humanized monoclonal antibody and Ang-2 antagonist peptide fusion protein, which has high specificity for the binding of VEGF-A and Ang-2.

SUMMARY:
The purpose of this Phase 1 study is comprised of multiple ascending-dose component (Part 1) and high concentration component (Part 2) to evaluate the safety, tolerability, pharmacokinetics, and efficacy of AM712 in patients with neovascular age- related macular degeneration (nAMD).

DETAILED DESCRIPTION:
The Part 1 of study is a multicenter, open-label, sequentially, multiple ascending-dose study to evaluate the safety, tolerability, pharmacokinetics, and efficacy of AM712 in subjects with nAMD.

Subjects will be sequentially enrolled into different dose-level cohorts following the traditional "3+3" design until the maximally tolerated dose (MTD) or the maximally administered dose (MAD) has been reached.

The Part 2 of study is a multicenter, open-label, sequential study to evaluate the safety, tolerability, pharmacokinetics, and efficacy of AM712 in treatment-naïve patients with nAMD.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects with 50 years of age or older
2. Active sub-foveal CNV lesion secondary to nAMD including juxta or extra-foveal lesions that partially affect the fovea
3. The area of CNV must occupy at least 50% of total lesion
4. Total lesion area ≤ 12 DA
5. ETDRS BCVA letter score measured at screening and baseline
6. Clear ocular media and adequate pupil dilation to permit good quality photographic imaging in study eye

Exclusion Criteria:

1. Any previous systemic anti-VEGF treatment
2. Any systemic treatment or therapy to treat neovascular AMD
3. Continuous use of systemic corticosteroids
4. Diseases that affect intravenous injection and venous blood sampling
5. Presence of CNV due to other causes, such as ocular histoplasmosis, trauma, multifocal choroiditis, angioid streaks, history of choroidal rupture, or pathologic myopia in study eye
6. History or any concurrent ocular condition which, in opinion of investigator, could either confound interpretation of efficacy and safety of IP or require medical or surgical intervention.
7. The area of fibrosis occupies ≥ 50% of total lesion area in study eye
8. Evidence of myopia degeneration, diagnosis supported by the axial length examination in study eye
9. History or any concurrent macular abnormality other than AMD in study eye
10. Current vitreous hemorrhage or history of vitreous hemorrhage in study eye
11. History of recurrent inflammation in study eye
12. History of treatment for nAMD
13. Subject having out of range laboratory values defined as:

ALT or AST > 2 x ULN, total bilirubin > 1.5 x ULN Serum creatinine > 1.5 x ULN, BUN > 2 x ULN HbA1c > 7.5% at screening

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2024-11-04 (Actual); Study Completion 2024-11-04 (Actual)

PRIMARY OUTCOMES:
Incidence of ocular adverse events (AEs) of the study eyes | 252 days
  To evaluate the safety and tolerability of AM712 in Subjects with neovascular Age-related Macular Degeneration (nAMD)
Incidence of non-ocular AEs | 252 days
  To evaluate the safety and tolerability of AM712 in Subjects with neovascular Age-related Macular Degeneration (nAMD)
Any relevant safety observations derived from BCVA | 252 days
  To evaluate the safety and tolerability of AM712 in Subjects with neovascular Age-related Macular Degeneration (nAMD)
Any relevant safety observations derived from SD-OCT | 252 days
  To evaluate the safety and tolerability of AM712 in Subjects with neovascular Age-related Macular Degeneration (nAMD)

SECONDARY OUTCOMES:
Mean change from baseline in central subfield thickness as assessed by SD-OCT | 252 days
  To evaluate the efficacy of AM712 in Subjects with nAMD
Proportion of patients with no intraretinal fluid, subretinal fluid, or pigment epithelial detachment as assessed by SD-OCT | 252 days
  To evaluate the efficacy of AM712 in Subjects with nAMD
Mean change from baseline in BCVA (ETDRS) | 252 days
  To evaluate the efficacy of AM712 in Subjects with nAMD
Proportion of patients gaining ≥ 15 letters from baseline BCVA | 252 days
  To evaluate the efficacy of AM712 in Subjects with nAMD

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Retina Consultants San Diego, Poway, California
  - Bay Area Retina Associates, Walnut Creek, California
  - Colorado Retina, Lakewood, Colorado
  - Florida Eye Associates, Melbourne, Florida
  - Retina Research Institute at New England Retina Consultants, Springfield, Massachusetts
  - Tennessee Retina, PC, Nashville, Tennessee
  - Retina Consultants of Texas, Bellaire, Texas
  - Retina Consultants of Texas, San Antonio, Texas
  - Retina Consultants of Texas, The Woodlands, Texas